CLINICAL TRIAL: NCT03230474
Title: Ultra Small Dose of Intrathecal Naloxone to Minimize Morphine Induced Side- Effects in Patients Undergoing Minor Anal Surgery Under Spinal Anesthesia. A Randomized Double Blind Study
Brief Title: a Small Dose of Naloxone,Minimize Intrathecal Morphine Side Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Lecturer of anesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00009914
Record Dates: First submitted 2017-07-23; First posted 2017-07-26 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Post-Op Complication
MeSH Terms: conditions — Postoperative Complications | interventions — Morphine; morphine 6-dehydrogenase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): 50 patients of this group will receive 5 mg of 0.5% hyperbaric bupivacaine with 0.2 mg morphine in 0.5 ml volume plus 0.5 ml as placebo (total volume 2 mL)
  Interventions: Drug: Morphine
- group 2 (Active Comparator): 50 patients of this group will receive 5 mg of 0.5% hyperbaric bupivacaine with 0.2 mg morphine in 0.5 ml volume plus 5ng\ kg naloxone in 0.5 ml volume (total volume 2mL).
  Interventions: Drug: Morphine-Naloxone

INTERVENTIONS:
Drug: Morphine — 50 patients of this group will receive 5 mg of 0.5% hyperbaric bupivacaine with 0.2 mg morphine in 0.5 ml volume plus 0.5 ml as placebo (total volume 2 mL)
  Arms: group 1
Drug: Morphine-Naloxone — 50 patients of this group will receive 5 mg of 0.5% hyperbaric bupivacaine with 0.2 mg morphine in 0.5 ml volume plus 5ng\ kg naloxone in 0.5 ml volume (total volume 2mL).
  Arms: group 2

SUMMARY:
I.V naloxone decreases incidence and severity of the common morphine side effects (pruritis, nausea/emesis, constipation, urinary retention, respiratory depression and undesirable sedation) so using it as additive to intrathecal morphine in patients undergoing anal surgeries under spinal anesthesia may be beneficail

DETAILED DESCRIPTION:
Bupivacaine hydrochloride is a commonly used local anesthetic in spinal anesthesia, however, the duration of spinal analgesia by bupivacaine is limited to about 75-150 minutes, therefore, various additives have been used along with bupivacaine for the prolongation of its effect, to improve the quality of analgesia, and to minimize the requirement for postoperative analgesics .

Opioids may be added to local anesthetic solutions to enhance surgical anesthesia and provide postoperative analgesia . This effect is mediated at the dorsal horn of the spinal cord, where opioids mimic the effect of endogenous enkephalins. The use of intrathecal (IT) morphine (0.1 to 0.5 mg) can provide effective control of postoperative pain for roughly 24 hours . However, the use of IT morphine may result in serious side effects e.g. pruritus 53%, nausea and vomiting 43%.urinary retention 43% and delayed respiratory depression . These side effects may lead to patient discomfort and prolonged hospital stay thus limiting the usefulness of IT morphine.

Naloxone has an extremely high affinity for μ-opioid receptors in the central nervous system (CNS). Naloxone is a μ-opioid receptor (MOR) competitive antagonist, and its rapid blockade of those receptors often produces rapid onset of withdrawal symptoms. Naloxone also has an antagonist action, though with a lower affinity, at κ- (KOR) and δ-opioid receptors (DOR). Unlike other opioid receptor antagonists, naloxone is essentially a pure antagonist with no agonist properties.

I.V naloxone decreases incidence and severity of the common morphine side effects (pruritis, nausea/emesis, constipation, urinary retention, respiratory depression and undesirable sedation) The addition of naloxone to morphine decreases the opioid related side effects without affection of postoperative analgesia. This combination can be used for the treatment of severe refractory chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I - II
* undergoing anal surgery with spinal anesthesia

Exclusion Criteria:

* Renal ,hepatic and cardiac patients -Infection at the site of injection.-
* Coagulopathy or other bleeding diathesis. -Preexisting neurologic deficits.-
* History of hypersensitivity to any of the given the drugs.
* Inability to communicate with the investigator and the hospital staff.
* History of chronic opioid use.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
post operative vomiting | 24 hours
  vomiting and nausea incidence

SECONDARY OUTCOMES:
pain | 24 hour postoperatively
  will be measured by VAS

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt